CLINICAL TRIAL: NCT07005115
Title: Analysis of Serum Lipid Profile in Patients With Lip Squamous Cell Carcinoma
Brief Title: Serum Lipid Profile and Lip Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alper Sindel, Professor, Akdeniz University
Other Study IDs: 22032023/250
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Lipid Profile; Lipids; SCC - Squamous Cell Carcinoma; Lip Cancer; Oral Cancer
Keywords: Oral Cancer; Lipids; Lipid Levels; Non-Smokers; Lip Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Lip Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: patients clinically evident and histopathologically confirmed with lip SCC
- control group: subjects without any underlying systemic disease

SUMMARY:
The goal of this observational retrospective study is to assess whether serum lipid levels differ between patients diagnosed with lip squamous cell carcinoma (SCC) and healthy individuals. The study aims to evaluate if alterations in lipid parameters, especially LDL levels, are associated with the presence of lip SCC and could serve as potential early biomarkers.

The main research questions are:

Do patients with lip SCC show significantly lower LDL levels compared to healthy controls? Are there significant differences in total cholesterol (TC), triglycerides (TG), HDL, and VLDL between the two groups? A retrospective analysis was conducted using existing medical records of patients with lip SCC and healthy subjects obtained from 2018-2023.

DETAILED DESCRIPTION:
Demographic data and lipid profile information were collected from 56 patients (28 lip SCC and 28 healthy). The lipid parameters included were total cholesterol (TC), triglycerides (TG), high density lipoprotein (HDL), low density lipoprotein (LDL) and very low-density lipoprotein (VLDL).

ELIGIBILITY:
Inclusion Criteria:

* patients clinically evident and histopathologically confirmed with lip SCC (study group)
* subjects without any underlying systemic disease (control group)

Exclusion Criteria:

* Age younger than 18 years
* pregnancy
* smoking
* history of radiotherapy or chemotherapy
* family history of hyperlipidemia
* accompanying malignancies other than lip SCC for both study and control groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data from patients with a histopathological diagnosis of primary lip cancers at Antalya Training and Research Hospital, Turkiye.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Low-Density Lipoprotein (LDL) Levels in Patients With Lip SCC vs. Healthy Controls | At time of diagnosis (retrospective data collection)
  To assess whether there is a statistically significant difference in fasting serum LDL levels between patients diagnosed with lip squamous cell carcinoma (SCC) and healthy subjects.

SECONDARY OUTCOMES:
Total Cholesterol (TC) Levels in Patients With Lip SCC vs. Healthy Controls | At time of diagnosis (retrospective data collection)
  To compare fasting serum total cholesterol (TC) levels between lip SCC patients and healthy controls.
Triglycerides (TG) Levels in Patients With Lip SCC vs. Healthy Controls | At time of diagnosis (retrospective data collection)
  To evaluate fasting serum TG levels in lip SCC patients compared to controls.
High-Density Lipoprotein (HDL) Levels in Patients With Lip SCC vs. Healthy Controls | At time of diagnosis (retrospective data collection)
  To compare HDL levels between lip SCC patients and healthy controls.
Very Low-Density Lipoprotein (VLDL) Levels in Patients With Lip SCC vs. Healthy Controls | At time of diagnosis (retrospective data collection)
  To compare fasting serum VLDL levels between study and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eldar Rasljanin, DDS, Principal Investigator — Akdeniz University, Antalya, Turkiye; Özer Erdem Gür, MD, Principal Investigator — Antalya Training and Research Hospital, University of Health Science, Antalya, Turkiye; Rezarta Taga Senirli, MD, Principal Investigator — Antalya Training and Research Hospital, University of Health Science, Antalya, Turkiye; Busehan Bilgin, DDS, Principal Investigator — Akdeniz University, Antalya, Turkiye; Öznur Özalp, DDS, Principal Investigator — Akdeniz University, Antalya, Turkiye; Mehmet Ali Altay, DDS, PhD, Principal Investigator — Akdeniz University, Antalya, Turkiye; Alper Sindel, DDS, PhD, Principal Investigator — Akdeniz University, Antalya, Turkiye
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lohe VK, Degwekar SS, Bhowate RR, Kadu RP, Dangore SB. Evaluation of correlation of serum lipid profile in patients with oral cancer and precancer and its association with tobacco abuse. J Oral Pathol Med. 2010 Feb;39(2):141-8. doi: 10.1111/j.1600-0714.2009.00828.x. Epub 2009 Dec 7. PMID 20002982
- [Background] Kark JD, Smith AH, Hames CG. Serum retinol and the inverse relationship between serum cholesterol and cancer. Br Med J (Clin Res Ed). 1982 Jan 16;284(6310):152-4. doi: 10.1136/bmj.284.6310.152. PMID 6799076
- [Background] Mehta R, Gurudath S, Dayansoor S, Pai A, Ganapathy KS. Serum lipid profile in patients with oral cancer and oral precancerous conditions. Dent Res J (Isfahan). 2014 May;11(3):345-50. doi: 10.4103/1735-3327.135889. PMID 25097644
- [Background] Kumar P, Augustine J, Urs AB, Arora S, Gupta S, Mohanty VR. Serum lipid profile in oral cancer and leukoplakia: correlation with tobacco abuse and histological grading. J Cancer Res Ther. 2012 Jul-Sep;8(3):384-8. doi: 10.4103/0973-1482.103517. PMID 23174719
- [Background] Gerber M, Richardson S, Crastes de Paulet P, Pujol H, Crastes de Paulet A. Relationship between vitamin E and polyunsaturated fatty acids in breast cancer. Nutritional and metabolic aspects. Cancer. 1989 Dec 1;64(11):2347-53. doi: 10.1002/1097-0142(19891201)64:113.0.co;2-v. PMID 2804926
- [Background] Forones NM, Falcao JB, Mattos D, Barone B. Cholesterolemia in colorectal cancer. Hepatogastroenterology. 1998 Sep-Oct;45(23):1531-4. PMID 9840100
- [Background] Neville BW, Day TA. Oral cancer and precancerous lesions. CA Cancer J Clin. 2002 Jul-Aug;52(4):195-215. doi: 10.3322/canjclin.52.4.195. PMID 12139232
- [Background] Patel PS, Shah MH, Jha FP, Raval GN, Rawal RM, Patel MM, Patel JB, Patel DD. Alterations in plasma lipid profile patterns in head and neck cancer and oral precancerous conditions. Indian J Cancer. 2004 Jan-Mar;41(1):25-31. PMID 15105576
- [Background] Alexopoulos CG, Blatsios B, Avgerinos A. Serum lipids and lipoprotein disorders in cancer patients. Cancer. 1987 Dec 15;60(12):3065-70. doi: 10.1002/1097-0142(19871215)60:123.0.co;2-q. PMID 3677028
- [Background] Acharya S, Rai P, Hallikeri K, Anehosur V, Kale J. Serum lipid profile in oral squamous cell carcinoma: alterations and association with some clinicopathological parameters and tobacco use. Int J Oral Maxillofac Surg. 2016 Jun;45(6):713-20. doi: 10.1016/j.ijom.2016.01.015. Epub 2016 Feb 19. PMID 26899131
- [Background] Bota JP, Lyons AB, Carroll BT. Squamous Cell Carcinoma of the Lip-A Review of Squamous Cell Carcinogenesis of the Mucosal and Cutaneous Junction. Dermatol Surg. 2017 Apr;43(4):494-506. doi: 10.1097/DSS.0000000000001020. PMID 28157733
- [Background] Moro JDS, Maroneze MC, Ardenghi TM, Barin LM, Danesi CC. Oral and oropharyngeal cancer: epidemiology and survival analysis. Einstein (Sao Paulo). 2018 Jun 7;16(2):eAO4248. doi: 10.1590/S1679-45082018AO4248. PMID 29898090
- [Background] Han AY, Kuan EC, Mallen-St Clair J, Alonso JE, Arshi A, St John MA. Epidemiology of Squamous Cell Carcinoma of the Lip in the United States: A Population-Based Cohort Analysis. JAMA Otolaryngol Head Neck Surg. 2016 Dec 1;142(12):1216-1223. doi: 10.1001/jamaoto.2016.3455. PMID 27832256
- [Background] Louredo BV, Vargas PA, Perez-de-Oliveira ME, Lopes MA, Kowalski LP, Curado MP. Epidemiology and survival outcomes of lip, oral cavity, and oropharyngeal squamous cell carcinoma in a southeast Brazilian population. Med Oral Patol Oral Cir Bucal. 2022 May 1;27(3):e274-e284. doi: 10.4317/medoral.25147. PMID 35368013
- [Background] Tranby EP, Heaton LJ, Tomar SL, Kelly AL, Fager GL, Backley M, Frantsve-Hawley J. Oral Cancer Prevalence, Mortality, and Costs in Medicaid and Commercial Insurance Claims Data. Cancer Epidemiol Biomarkers Prev. 2022 Sep 2;31(9):1849-1857. doi: 10.1158/1055-9965.EPI-22-0114. PMID 35732291